CLINICAL TRIAL: NCT01840514
Title: Cardiac Functions in Living Donor Liver Transplant Recipients. An Echocardiographic Study.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amr Mohamed Yassen, professor, Mansoura University
Other Study IDs: 1982
Record Dates: First submitted 2013-04-23; First posted 2013-04-25 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: Liver Transplant
Keywords: recipient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day

SUMMARY:
The stress of orthotopic living donor liver transplantation in patients with cirrhosis could induce worsening of an already recorded myocardial dysfunction or may be associated with a new myocardial dysfunction in patients previously having normal myocardial functions, therefore this study will be designed for intra-operative detection of new onset ventricular dysfunction or worsening of already diagnosed ventricular dysfunction in living donor liver transplant recipient and the possible contribution of several hemodynamic and oxygenation parameters in the generation of any cardiovascular function impairment will be also investigated and to determine the impact of ventricular dysfunction on early (7 PO days) graft function, 28 days survival and patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* all adult recipient

Exclusion Criteria:

* massive blood transfusion
* grade III esophageal varices

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: recipient of living donor liver
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2012-12; Primary Completion 2015-04 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
hemodynamic monitoring | intraoperative

SECONDARY OUTCOMES:
graft function | 7 days

OTHER OUTCOMES:
survival | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: amr yassen, MD, Principal Investigator — Liver transplant program, mansoura faculty of medicine
Locations (2):
- Egypt (2):
  - Liver transplantation program - Gastroenterology surgical center, Al Mansurah, Dakahlia Governorate
  - Liver transplantation project - Gastroenterology surgical center - Mansoura university, Al Mansurah, Dakahlia Governorate